CLINICAL TRIAL: NCT02261389
Title: Three-monthly Dynamic Evaluation of CEA and CA 15.3 vs Usual Practice in the Follow-up of Early Breast Cancer Patients: a Randomized Study
Brief Title: Follow-up of Early Breast Cancer by Dynamic Evaluation of CEA and CA 15.3 Followed by 18FDG-PET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: PONS-S (Patientenorientierte Nachsorge-Stiftung), Augsburg, Germany (Unknown); Azienda ULSS 12 Veneziana (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Claudio Zamagni MD, MD Medical Oncologist, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KRONOS; PONS-S Italy (Other: S.Orsola-Malpighi Hospital)
Record Dates: First submitted 2014-09-30; First posted 2014-10-10 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; follow-up; tumor markers
MeSH Terms: conditions — Breast Neoplasms | interventions — Mucin-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A, usual follow-up practice (No Intervention): Imaging studies and serum markers (CEA, CA 15.3, others) performed according to local practice
- Arm B, tumor markers assessment (Experimental): Serum CEA and CA 15.3 performed every 3 months. No imaging studies allowed in asymptomatic patients: imaging studies (18 FDG-PET) performed only in case of critical increase of CEA and /or CA 15.3 serum levels (+100% for CEA and +75% for CA15.3), even if in the normal range.
  Interventions: Other: Arm B, tumor markers assessment

INTERVENTIONS:
Other: Arm B, tumor markers assessment — Tumor markers assessment every three months through the study or until disease recurrence
  Other Names: CEA; CA15-3; 18FDG-PET
  Arms: Arm B, tumor markers assessment

SUMMARY:
The main purpose of follow-up in asymptomatic breast cancer patients during and after adjuvant treatment is to detect breast cancer recurrence and metastatic disease.The aim of this trial is to verify if, in asymptomatic patients, the serial measurement of serum CEA and CA 15.3, with diagnostic imaging procedures (18FDG-PET) performed only in case of a critical increase of serum CEA and CA 15.3 level, can anticipate the diagnosis of breast cancer local and distant recurrence compared to the usual follow-up practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years.
* Histologically confirmed stage I-III epithelial breast cancer.
* Adequate surgery of breast and axilla:

  1. patients must have undergone either a total mastectomy or breast conserving surgery
  2. surgical margins of the resected specimen must be histologically free of invasive tumor.
* Cohort 1: if chemotherapy and/or radiotherapy are indicated the patients must be randomized between 1 month and 2 months from the end of chemotherapy and/or radiotherapy; if only hormonal adjuvant therapy is indicated the patients must be randomized within 3 months from the completion of surgery
* Cohort 2: patients must be randomized in the trial after 5 years of follow-up without relapse (but within year 6)
* Signed informed consent obtained prior to any study-specific procedures.

Exclusion Criteria:

* Histologically confirmed stage 0 epithelial breast cancer (carcinoma in situ).
* Special histologies with a high or low risk of relapse (i.e. sarcoma and tubular carcinoma)
* T1a and T1b tumors with all the following characteristics: G1-2 and N0 and RE > 10%, RPg > 10% and HER2 negative and Ki67≤14%
* Evidence of distant metastases
* Patients participating to other clinical trials requiring follow-up not equal to standard
* Previous history of cancer within 5 years from randomization (except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, stage I uterine cancer, or other non-breast malignancies with an outcome similar to those mentioned above)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1507 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Time interval between date of randomization and date of diagnosis of disease distant recurrence | Participants will be followed from date of randomization until the date of first documented disease distant recurrence or date of death from any cause, whichever came first, assessed up to 60 months
  Primary objective of the study is to verify if the experimental arm (serial measurement of serum CEA and CA 15.3 with diagnostic imaging procedures - i.e. 18FDG-PET- performed only in case of critical increase of serum markers level) can anticipate the diagnosis of breast cancer loco-regional (except for in-breast recurrence) or distant metastases compared to the control arm (usual follow-up practice).

SECONDARY OUTCOMES:
Predefined critical difference of CEA and CA15-3 | Participants will be followed from date of randomization until the date of first documented disease distant recurrence or date of death from any cause, whichever came first, assessed up to 60 months
  Secondary objective is to evaluate the Positive Predictive Value (PPV) and the Negative Predictive Value (NPV) of CEA and CA15.3 dynamic changes in the diagnosis of breast cancer loco-regional (except for in-breast recurrence) or distant metastases.
Exploratory analysis in the different subtypes | Participants will be followed from date of randomization until the date of first documented disease distant recurrence or date of death from any cause, whichever came first, assessed up to 60 months
  Secondary objective is to perform an exploratory analysis on diagnostic anticipation in the different subtypes (ER and HER2 status)
Imaging diagnostic tests evaluation | Participants will be followed from date of randomization until the date of first documented disease distant recurrence or date of death from any cause, whichever came first, assessed up to 60 months
  Secondary objective is to measure how many imaging diagnostic tests will be avoided in the experimental arm compared to the control arm
Patient quality of life evaluation | Participants will be followed from date of randomization until the date of first documented disease distant recurrence or date of death from any cause, whichever came first, assessed up to 60 months
  Secondary objective is to compare the quality of life in the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Zamagni, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Bologna
Locations (7):
- Italy (7):
  - Azienda Sanitaria dell'Alto Adige - Ospedale di Bressanone, Brixen, Bolzano
  - Azienda Sanitaria dell'Alto Adige - Ospedale di Merano, Merano, Bolzano
  - ASL13 - Presidio Ospedaliero Mirano, U.O.C. Oncologia ed Ematologia Oncologica, Mirano, Venezia
  - Azienda Ospedaliero-Universitaria di Bologna, Policlinico S. Orsola-Malpighi, SSD Oncologia Medica Addarii, Bologna
  - Azienda Sanitaria dell'Alto Adige - Ospedale Centrale di Bolzano, Bolzano
  - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara
  - IRCCS Azienda Ospedaliera S. Maria Nuova di Reggio Emilia, Reggio Emilia